CLINICAL TRIAL: NCT04933396
Title: Accuracy of the Recent Consensus Based Definition of FGR Encompassing Biometric and Doppler Parameters in Predicting Adverse Neonatal Outcomes
Brief Title: FGR Diagnostic Criteria in Predicting Adverse Neonatal Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, associate professor, Ain Shams University
Other Study IDs: Asu FM
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: FGR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound diagnostic criteria — evaluate using the recent consensus based definition for FGR using biometric and Doppler parameters to identify fetuses at risk of adverse perinatal outcomes compared to using solely biometric based parameter (EFW <10th percentile according to the Hadlock growth standard).

SUMMARY:
The purpose of this study is to evaluate using the recent consensus based definition for FGR using biometric and Doppler parameters to identify fetuses at risk of adverse perinatal outcomes compared to using solely biometric based parameter (EFW <10th percentile according to the Hadlock growth standard).

ELIGIBILITY:
Inclusion Criteria:

* Participants included in this study will have the following criteria:

  * Pregnancies complicated with FGR (EFW <10th percentile).
  * Singleton pregnancy.

Exclusion Criteria:

* • Fetal structural malformations or chromosomal abnormalities as detected by neonatal examination and anomaly scan during pregnancy.

  * Identified infectious etiologies detected during immediate postnatal examination or during pregnancy.
  * Gestational age cannot be calculated accurately.
  * Missing antenatal or perinatal outcome data.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all pregnancies with FGR (EFW <10th percentile) who were admitted in Ain Shams University Maternity Hospital during the period from January 2016 till December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
adverse events | 30 days after delivery
  neonatal outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No